CLINICAL TRIAL: NCT05223257
Title: Action Observation Tele-rehabilitation for Upper Limb in Children With Diplegic Cerebral Palsy
Brief Title: Action Observation in Children With Diplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: IRCCS reggio emilia (Unknown); University of Parma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2019-12370746
Record Dates: First submitted 2021-12-17; First posted 2022-02-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Tele-rehabilitation; Action Observation; Mirror neurons; ICT
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be a parallel RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): AOT is based on the observation of meaningful actions followed by their execution
  Interventions: Other: AOT
- Control group (No Intervention): Children will continue standard care for 8 weeks
  Subject allocated to "standard care" group will have to continue what they normally do; they (if > 13 years) or their parents will have to fill a diary in which they will write the rehabilitative activities they do, specifying their intensity and whether these activities are more focused on the lower limbs or upper limbs.

INTERVENTIONS:
Other: AOT — Observation of video sequences showing unimanual and bimanual goal-directed actions followed by the execution of the observed actions with upper limbs for unimanual and bimanual actions.
  Arms: Experimental group

SUMMARY:
A new rehabilitative approach, called AOT, based on the discovery of mirror neuron system (MNS), has been used with promising results on the Upper Limb (UL) function in some studies in children with Cerebral Palsy (CP).

The purpose of the present trial is to provide evidence by an RCT, preceded by a pilot study, that customized and home based AOT training is an effective rehabilitation tool in children with diplegic CP (DCP) and that its effects are greater than standard care.

Both Hands Assessment (BoHA) is chosen as primary outcome measure and a sample size of 27 per group is required. The rehabilitation lasting 8 weeks will be provided at home by an ICT platform able to deliver, manage, monitor and measure a personalized AOT.

DETAILED DESCRIPTION:
A two-arm, evaluator-blinded, randomized trial (RCT), preceded by a pilot study, will be conducted according to CONSORT guidelines. Each participant will be randomized to either:

1. Intervention group (Experimental group). Children will receive immediately the system for 8 weeks.
2. Standard care group (Control group). Children will continue standard care At the end of the project, if the study results will be positive, children enrolled in the control group will be able to have the same treatment as the experimental group, if necessary.

The system will provide an in-home, individualized, intensive treatment based on the AOT. The system will be delivered at home and the children will perform a 60-minute training session at least 5 days a week for 8 consecutive weeks (total of 40 hours).

Follow-up assessment (outcome measures) will be conducted before (T0) and post-intervention at 1 weeks (T1), and then 8 and 24 weeks after the AOT intervention/standard care (T2 and T3).

The primary endpoint will be T1. Clinical assessments will be administered by a therapist blind to group assignment in each centre. Scoring of videotaped clinical outcome measures will be performed by therapists blind to group allocation and assessment order.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diplegic cerebral palsy (DCP) (GMFCS level I to IV - children may have been achieved an independent gait)
* age between 5 and 16 years
* MACS level I-IV
* sufficient cooperation and communicative understanding to perform assessments and participate in the intervention
* caregivers able to commit and collaborate in a rehabilitative intensive home
* subjects and parents able to commit to the intensive rehabilitation program for a period of 8 weeks.

Exclusion Criteria:

* Exclusion criteria will be uncontrolled seizures and UL botulinum injections or orthopaedic surgery in the previous 6 months or during the study period.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-09-16 (Estimated)

PRIMARY OUTCOMES:
Changes in the Both Hands Assessment (BoHA) | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  This assessment measures bimanual performance in children with bilateral CP, during a semi-structured session with specific toys or activities.

SECONDARY OUTCOMES:
Changes in Melbourne Assessment 2 (MA2) | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  It is criterion-referenced test that measures unilateral upper extremity quality of movement in subjects with neurological impairments.
Changes in Box and Block Test (BBT) | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  It measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations from childhood to adults.
Changes in cognitive assessment | Baseline (T0, 1 week before beginning of the study)
  It will be done cognitive assessment with the Wechsler Intelligence Scale for Children (WISC) that is an individually administered intelligence test for children.
Changes in neuropsychological assessment (social perception domain) | Baseline (T0, 1 week before beginning of the study)
  It will be done neuropsychological assessment with NEPSY-2 social perception domains, that measures the ability to: understand social contexts, interpret non verbal communication, form impressions of others, use contextual information to make inferences about others and their behaviour.
Changes in neuropsychological assessment (sensory-motor domain) | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period); T3 (24 weeks after the end of the training/control period)
  It will be done neuropsychological assessment with NEPSY-2 sensory-motor domains, that consists of four tests that evaluate motor speed and precision, the ability to plan and execute movement sequences, bimanual and visuomotor coordination and imitation of movement.
Changes in BRIEF P | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period); T3 (24 weeks after the end of the training/control period)
  The Behavior Rating Inventory of Executive Function (BRIEF) measures the executive function in daily life context of children from the parents point of view. BRIEF P is for pre-school children.
Changes in BRIEF 2 | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period); T3 (24 weeks after the end of the training/control period)
  The Behavior Rating Inventory of Executive Function (BRIEF) measures the executive function in daily life context of children from the parents point of view. BRIEF 2 is for school children.
Changes in ABILHAND-kids | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  A semi-structured item-response questionnaire that measures manual ability according to a caregiver's perceived difficulty performing daily bimanual tasks.
Changes in Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL -Child, 4-12 years) | Baseline (T0) and T3 (24 weeks after the end of the training/control period)
  This instrument is useful for evaluating interventions designed to improve the lives of children.
Changes in Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL -Teen, 13-18 years) | Baseline (T0) and T3 (24 weeks after the end of the training/control period)
  This instrument is useful for evaluating interventions designed to improve the lives of adolescents.
Changes in Participation and Environment Measure - Children and Youth (PEM-CY) | Baseline (T0) and T3 (16 weeks after T2)
  It is a measure that evaluates participation in the home, at school, and in the community, alongside environmental factors within each of these settings.
Changes in Canadian occupational performance measure (COPM) | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  It is a validated measure that aims to identify rehabilitation needs in daily life and changes by the subject or his family.
Changes in technological measurement of manual abilities by means of Virtual Reality Rehabilitation System (VRRS) | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  VRRS activities are aimed at estimating and evaluating the uni and bimanual activities, quantitatively through kinematic parameters.
Changes in technological measurement of manual abilities by means of Upper Limb TRAcker system (ULTRA +) | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  ULTRA+ is a sensorized biomechatronic system equipped with an articulated arm with seven degrees of freedom. Kinematic and grip strength parameters will be obtained, thanks to a real immersion in a three-dimensional virtual environment.
Feasibility questionnaire | T1 (within 1 week after the end of the training)
  In order to investigate the feasibility of the system and the compliance of children and their families, will be carried out a questionnaire ad hoc at the end of the T1 assessment training in the experimental group.
Changes in cerebral plasticity with fMRI (Functional Magnetic Resonance Imaging) | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period)
  A subgroup of children, selected based on specific inclusion sub-criteria, will be asked to perform the fMRI examination before (T0) and immediately after the end of the experimental or standard treatment period (T1). The children will perform two tasks:
  1. Motor execution
  2. Action observation task In order to understand the feasibility of these tasks and the brain circuits involved during their execution, a group of typically developing children and healthy young adults will also be enrolled on a voluntary basis.
  The fMRI study will evaluate the difference in intensity and extension of brain activation in relation to the rehabilitation intervention, as well as to demonstrate the effectiveness of the experimental rehabilitation intervention compared to the control one.
Quantitative Changes in upper limbs activities detected with Actigraph GXT3+ during clinical assessment. | Baseline (T0, 1week before beginning of the study); T1 (within 1 week after the end of the training/control period); T2 (8 weeks after the end of the training/control period) and T3 (24 weeks after the end of the training/control period)
  Actigraph GXT3+ worn during BoHA assessments
Changes in daily life activities detected with Actigraph GXT3+ | During training and/or standard period (from T0 to T1) (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the training/control period)
  Quantitative measurement of daily manual activities

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - University of Parma, Parma
  - IRCCS Fondazione Stella Maris, Pisa
  - IRCCS Reggio Emilia, Reggio Emilia

REFERENCES:
- [Background] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Biagi L, Tosetti M, Fogassi L, Cioni G. Upper limb children action-observation training (UP-CAT): a randomised controlled trial in hemiplegic cerebral palsy. BMC Neurol. 2011 Jun 28;11:80. doi: 10.1186/1471-2377-11-80. PMID 21711525
- [Background] Buchignani B, Beani E, Pomeroy V, Iacono O, Sicola E, Perazza S, Bieber E, Feys H, Klingels K, Cioni G, Sgandurra G. Action observation training for rehabilitation in brain injuries: a systematic review and meta-analysis. BMC Neurol. 2019 Dec 27;19(1):344. doi: 10.1186/s12883-019-1533-x. PMID 31881854
- [Background] Sgandurra G, Cecchi F, Beani E, Mannari I, Maselli M, Falotico FP, Inguaggiato E, Perazza S, Sicola E, Feys H, Klingels K, Ferrari A, Dario P, Boyd RN, Cioni G. Tele-UPCAT: study protocol of a randomised controlled trial of a home-based Tele-monitored UPper limb Children Action observation Training for participants with unilateral cerebral palsy. BMJ Open. 2018 May 14;8(5):e017819. doi: 10.1136/bmjopen-2017-017819. PMID 29764869
- [Background] Beani E, Menici V, Ferrari A, Cioni G, Sgandurra G. Feasibility of a Home-Based Action Observation Training for Children With Unilateral Cerebral Palsy: An Explorative Study. Front Neurol. 2020 Feb 28;11:16. doi: 10.3389/fneur.2020.00016. eCollection 2020. PMID 32180754
- [Background] Sgandurra G, Biagi L, Fogassi L, Ferrari A, Sicola E, Guzzetta A, Tosetti M, Cioni G. Reorganization of action observation and sensory-motor networks after action observation therapy in children with congenital hemiplegia: A pilot study. Dev Neurobiol. 2020 Sep;80(9-10):351-360. doi: 10.1002/dneu.22783. Epub 2020 Oct 28. PMID 32986904